CLINICAL TRIAL: NCT02477852
Title: The Study of Standardized Preoperative Anti-tuberculosis Treatment of Surgical Treatment of Spinal Tuberculosis Patients
Brief Title: The Optimal Duration of Preoperative Anti-tuberculosis Treatment of Spinal Tuberculosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Jing Liu, Administrator, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D141107005214002
Record Dates: First submitted 2015-05-23; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Tuberculosis, Spinal
Keywords: tuberculosis; spinal; general; operation; drug; therapy
MeSH Terms: conditions — Tuberculosis, Spinal; Tuberculosis | interventions — Isoniazid; Rifampin; Ethambutol; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anti-tuberculosis treatment two weeks (Experimental): anti-tuberculosis drugs All the patients in the groups receive anti-tuberculosis treatment with Isoniazid 0.3g po qd, Rifampicin 0.45g po qd, Ethambutol 0.75 g po qd,Pyrazinamide 0.5g po tid. for two weeks.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Ethambutol; Drug: Pyrazinamide
- anti-tuberculosis treatment four weeks (Experimental): anti-tuberculosis drugs All the patients in the groups receive anti-tuberculosis treatment with Isoniazid 0.3g po qd, Rifampicin 0.45g po qd, Ethambutol 0.75 g po qd,Pyrazinamide 0.5g po tid. for four weeks.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Ethambutol; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Isoniazid — preoperative treatment of spinal tuberculosis with Isoniazid
Drug: Rifampicin — preoperative treatment of spinal tuberculosis with Rifampicin
Drug: Ethambutol — preoperative treatment of spinal tuberculosis with Ethambutol
Drug: Pyrazinamide — preoperative treatment of spinal tuberculosis with Pyrazinamide

SUMMARY:
The purpose of this study is to determine the better preoperative anti-tuberculosis treatment period of patients with spinal tuberculosis.

DETAILED DESCRIPTION:
Quality assurance plan：All the investigators will receive uniform training. Standard cases follow-up,collection,management systems will be established.The process of cases follow-up,collection,management will be supervised by the third party.Data entry will be in the manner of independent parallel entry.The endpoints events are judged by third party.Statistical analysis are implemented by the statistics institutions of the third party.In order to control the bias,this study takes multicenter,random,control study design.

Sample size assessment:Under the condition of multicenter,random,control design, computational formula takes the rate comparisons of two groups.The key endpoints event is soft tissue width of vertebral side measured by computed tomography. The incidence of the key endpoints event in two weeks group is 30%.The incidence of the key endpoints event in four weeks group is 15%.When alpha value is 0.5 and power value is 0.9,the sample size is 161 patients.If loses visit rate is 20%,the sample size is 194 patients.

Statistical analysis plan:The key events are analyzed by chi-squared test.The statistical significance factors among them are calculated by relative risk.

Data checks and source data verification are supervised by a third-party organization (contract research organization，CRO).

Standard Operating Procedures:Investigator's brochure has explained in detail about the standard operating procedures of everything.Data dictionary can be found in standard operating procedures.

Plan for missing data: The investigators Set a 20% rate of lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed as spinal tuberculosis clinically,and they do not receive antituberculosis therapy or with 2 weeks.
* The age is between 15 years old and 75 years old.
* Patients have good compliance,and have clear surgical indications.4.Willing to join the research

Exclusion Criteria:

* Patients have surgical contraindications.
* Patients have bad habits:taking drug,drinking.3.Patients have mental disease.
* Patients have bad compliance.
* Patients have hematogenous disseminated pulmonary tuberculosis, serious central nervous system tuberculosis,and serious extrapulmonary tuberculosis.
* Patients with drug resistance for Antituberculosis drugs,and patient have to change the treat plan,and patients have immunodeficiency diseases.
* Patients are not diagnosed as spinal tuberculosis clearly.
* Not willing to join the research

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Vertebral side width of soft tissue is measured by CT after operation. | up to 3 months

SECONDARY OUTCOMES:
Amount of bone trabecula between bone graft surfaces is measured by X-ray after operation. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: shao fa xu, doctor, Study Chair — Beijing Chest Hospital
Locations (1):
- Beijing chest hospital, Beijing, Beijing Municipality, China